CLINICAL TRIAL: NCT02046330
Title: Deep Brain Stimulation (DBS) Therapy for Treatment Resistant
Brief Title: Deep Brain Stimulation (DBS) Therapy for Treatment Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jair Soares, Professor and Chair, Psy-Behavioral Sciences, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-13-0004
Record Dates: First submitted 2013-12-17; First posted 2014-01-27 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
Keywords: Deep Brain Stimulation; Treatment Resistant Depression; Major Depressive Disorder; Depression; ECT; TNS
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): Device implantation (Deep Brain Stimulation Model 3387 Model 3389)
  Interventions: Device: Deep Brain Stimulation Model 3387 Model 3389

INTERVENTIONS:
Device: Deep Brain Stimulation Model 3387 Model 3389 — Implantation of all devices will be performed at a single session. Lead implantation will take place under local anesthesia, with implanted pulse generator (IPG) implantation under general anesthesia. The stereotaxic frame will be fitted on the day of surgery, following standard stereotactic surgical procedure. The leads will be inserted so that the stimulation sites span superolateral median forebrain bundle.
  Other Names: Medtronic Neuromodulation

SUMMARY:
We propose a clinical study of medial forebrain bundle DBS as a treatment in 20 patients with treatment refractory depression (TRD). Data from the University of Bonn indicates that surgical lesions of the medical forebrain bundle can produce therapeutic benefits in patients with depressive disorders, and suggest that DBS at the same site may also reduce symptomatology in these TRD patients (Schaepfer, 2013). Depression affects up to 10% of the US population and of those at least 10-15% do not benefit from therapies hence why we must explore new treatments. The Percept™ PC system manufactured by Medtronic Neurological will be used in this study. Study subjects will be between the ages of 22 and 70 years of age and suffer from TRD, have failed multiple treatment regimens, including ECT, and remain symptomatic. Those identified as TRD patients will then be enrolled in a clinical pilot study investigating DBS, targeting the MFB.

DETAILED DESCRIPTION:
Study Design: Subjects will be ten patients with MDD identified via the Structured Clinical Interview for DSM-IV, manifesting a current major depressive episode of disabling severity, refractory to prolonged treatment trials with conventional medication, electro-convulsive therapy (ECT) and psychotherapy. A marked impact of depression on their health and functional status will be evidenced by major impairment in functioning or potentially severe medical outcomes (repeated hospitalizations, serious suicidal or other self-injurious behavior). They will be recruited from individuals currently seen at our facility or referred by psychiatrists in the community. Patients will be initially screened by a comprehensive review of their psychiatric history, obtained by interview of the patient, family and treating psychiatrist and/or psychologist, as well as by obtaining and reviewing all available records of previous psychiatric treatment. The available generally-accepted alternative treatments for depression are pharmacologic therapy, psychotherapy, and ECT. Failed trials of multiple proven pharmacologic treatments, an adequate course of psychotherapy, and an adequate course of bilateral ECT (or inability to tolerate an adequate ECT trial) are inclusion criteria for all candidates who are considered for this study. However, as alternatives to participation in this study, candidates may undertake additional trials of potentially beneficial novel combinations of medication and psychotherapy, or they may undertake trials of novel interventions lacking definitive evidence of efficacy in severe depression (e.g., light therapy, herbal therapy, transcranial magnetic stimulation, vagal nerve stimulation). The protocol was designed to include four phases. All patients will enter these phases in the same sequence. The experimental design is illustrated in the timeline in Figure 1. Surgical implantation will be followed by: 1) Baseline Phase (a 1 month period with no stimulation); 2) Variable Staggered Phase (blinded stimulation onset starting from 1 month to 3 months post implant, with optimal parameter determination during this time ; 3) Initial Chronic Phase (blinded bilateral stimulation, lasting at least three months) (see below); 4) Continuation Phase (unblinded active bilateral or unilateral stimulation to maximize clinical response) Protocol overview and design: We propose a clinical study of medial forebrain bundle DBS as a treatment in 10 patients with treatment refractory depression (TRD). Data from the University of Bonn indicates that surgical lesions of the medical forebrain bundle can produce therapeutic benefits in patients with depressive disorders, and suggest that DBS at the same site may also reduce symptomatology in these TRD patients (Schaepfer, 2013). Depression affects up to 10% of the US population and of those at least 10-15% do not benefit from therapies hence why we must explore new treatments. The Percept™ PC system manufactured by Medtronic Neurological will be used in this study. Those identified as TRD patients will then be enrolled in a clinical pilot study investigating DBS, targeting the MFB.

ELIGIBILITY:
Inclusion Criteria:

1. Major Depression Disorder (MDD) diagnosed by Structured Clinical Interview for DSM-IV (SCID I/DSM-IV), judged to be of disabling severity.
2. Age 22 - 70 years.
3. 24-item Hamilton Depression Rating Scale (HDRS) score of at least 21 on the first 17 items
4. Global Assessment of Function (GAF) score of 45 or less.
5. A recurrent (equal or >4 episodes) or chronic (episode duration equal or higher >2 years) course AND a minimum of 5 years since the onset of the first depressive episode. Major impairment in functioning or potentially severe medical outcomes (repeated hospitalizations, serious suicidal or other self-injurious behavior).
6. Failure to respond to: 6.1. Adequate trials (equal or >6 weeks at the maximum recommended or tolerated dose) of primary antidepressants from at least 3 different classes AND; 6.2. adequate trials ( equal>4 weeks at the usually recommended or maximum tolerated dose) of augmentation/combination of a primary antidepressant using at least 2 different augmenting/combination agents (lithium, T3, stimulants, neuroleptics, anticonvulsants, buspirone, or a second primary antidepressant) AND; 6.3 An adequate trial of ECT (>6 bilateral treatments), or inability to tolerate an adequate ECT trial, AND; 6.4 An adequate trial of individual psychotherapy (>20 sessions with an experienced psychotherapist).
7. Able to comply with the operational and administrative requirements of participation in the study.
8. Able to give written informed consent
9. On a stable drug regimen of psychotropic medication for at least 6 weeks at the time of entry into the study.
10. Good general health. No changes in medication treatment during participation in study.

Exclusion Criteria:

1. Current or past non-affective psychotic disorder, Bipolar Disorder, Schizophrenia, or Schizoaffective disorder. Patients who suffer from generalized anxiety disorder will be permitted to participate as long as MDD is the primary clinical diagnosis.
2. Any current clinically significant neurological disorder, including dementia or medical illness affecting brain function.
3. Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI).
4. Any previous surgery to destroy the region of the brain that will be the target of treatment.
5. Any surgical contraindications to undergoing DBS, including labeled contraindications for DBS and/or inability to undergo presurgical MRI (cardiac pacemaker, implantable defibrillator or other implantable stimulator, pregnancy, metal in body, severe claustrophobia), infection, coagulopathy, inability to undergo an awake operation, significant cardiac or other medical risk factors for surgery.
6. Refusal of an adequate trial of ECT.
7. History of stimulation intolerance in any area of the body.
8. Current or unstably remitted substance abuse or dependence. No alcohol and/or substance abuse or dependence in the past 6 months.
9. Pregnancy and women of childbearing age not using effective contraception. Double-barrier method is required.
10. History of severe personality disorder, where, based on the judgment of the investigators, the personality disorder will interfere with the patient's ability to complete the follow-up protocol, e.g. borderline personality disorder.
11. Imminent risk of suicide
12. Participation in another drug, device, or biologics trial within the preceding 30 days
13. Presence of a condition requiring routine MRIs.
14. Presence of a condition requiring diathermy.
15. Subject is on anticoagulant medication.
16. Not able to comply with the operational and administrative requirements of participation in the study (based on the judgment of the investigators).
17. Terminal illness associated with expected survival of <12 months.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-12-16 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes in patients MADRS scores | weekly (24 Months)
  We will assess individual patient response, measured by standardized patient and clinician ratings of depression severity, under blinded conditions. Prospective ratings using validated and reliable measures of symptoms, quality of life and safety will be employed. We will assess safety for all subjects by monitoring any adverse events.

SECONDARY OUTCOMES:
Accuracy of Electrode placement | Post-operation (weekly for 24 months)
  We will implant the Model 3387/Model 3389 lead at this target location, with the exact choice of lead to be determined during surgery.
Frequency and Charge of Stimulation | Weekly (24 months total)
  The optimal stimulation parameters for reducing depressive symptoms acutely and chronically are unknown. Preliminary data suggest that psychiatric patients who have responded to DBS have responded at high frequencies and amplitudes that presumably induce a depolarization block or "neuronal jamming," and thus mimic a lesion. We intend to explore the effects of a wide range of frequencies and amplitudes during the acute testing phase and to utilize high frequency continuous stimulation at the lowest amplitude that results in a definitive effect in the chronic phase of the study.
Determine Feasibility of a Double Blind Study | 24 months
  We hypothesize that it will be possible to develop a suitable double-blind procedure by which neither patients nor physicians will know whether DBS is on or off at any given moment.
Decrease in Neurocognitive scores on CSTC | pre-operative, 12 month and 24 months post-operation
  In this study, neuropsychological tests believed sensitive to changes in Concept Shifting Test-Combined (CSTC) function, and particularly orbitofrontal function, will be obtained with the stimulator on and off, if possible, under blinded conditions. In a separate study, positron emission tomography (PET) perfusion imaging and neuropsychological tests will be obtained to determine how corticobasal brain function changes after acute and chronic DBS.
Assess maintenance of treatment response (or remission) associated with chronic DBS: | 6, 12, and 24 months
  Maintaining Treatment Response
Number of Adverse Events | 24 months (reported weekly)

CONTACTS AND LOCATIONS:
Overall Officials: Jair C Soares, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Joao Quevedo, MD, PhD, Study Director — The University of Texas Health Science Center, Houston; Giovana Zunta Soares, MD, Study Director — The University of Texas Health Science Center, Houston
Locations (1):
- UT Center of Excellence on Mood Disorders, Houston, Texas, United States

REFERENCES:
- [Derived] Fenoy AJ, Schulz P, Selvaraj S, Burrows C, Spiker D, Cao B, Zunta-Soares G, Gajwani P, Quevedo J, Soares J. Deep brain stimulation of the medial forebrain bundle: Distinctive responses in resistant depression. J Affect Disord. 2016 Oct;203:143-151. doi: 10.1016/j.jad.2016.05.064. Epub 2016 Jun 3. PMID 27288959